CLINICAL TRIAL: NCT00969384
Title: Physical Health of Residents in Psychiatric Institutions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Enheden for psykiatrisk forskning, Region Nordjylland
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3,3 270809
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2009-09-01 (Estimated); Status verified 2009-08

CONDITIONS: Physical Health
Keywords: Physical health; Mental illness; prevention; Waist circumference
MeSH Terms: conditions — Mental Disorders

ARMS (2):
- waist circumferences (Experimental): Intervention (active awareness):
  In the intervention institutions, a detailed feedback of all index measures will be distributed to the patients and the staff. The project leader and a medical specialist in psychiatry will advise on medical aspects and health promotion. In connection with this feedback, guidance on psycho-pharmacological treatment will be provided.
  Interventions: Behavioral: Active awareness/Lifestyle counseling
- Lifestyle counseling (Experimental): Intervention (active awareness):
  In the intervention institutions, a detailed feedback of all index measures will be distributed to the patients and the staff. The project leader and a medical specialist in psychiatry will advise on medical aspects and health promotion. In connection with this feedback, guidance on psycho-pharmacological treatment will be provided.
  Interventions: Behavioral: Active awareness/Lifestyle counseling

INTERVENTIONS:
Behavioral: Active awareness/Lifestyle counseling — Intervention (active awareness):
  In the intervention institutions, a detailed feedback of all index measures will be distributed to the patients and the staff. The project leader and a medical specialist in psychiatry will advise on medical aspects and health promotion. In connection with this feedback, guidance on psycho-pharmacological treatment will be provided.

SUMMARY:
Aim of the study: To investigate if the intervention described in this protocol has an effect on patients' and staff's physical health.

Null hypothesis: There is no difference in waist circumference, body weight, quality of life and the rate of polypharmacy between the intervention and control groups after six months.

DETAILED DESCRIPTION:
Background:

The prevalence of physical health problems among patients suffering from psychiatric illnesses is above that seen in the average population (1). Cardiovascular diseases (2) and metabolic disorders (3;4) are common in persons diagnosed with schizophrenia (5;6). A fact that has been known for many years (7), and there has been no decrease in the prevalence of physical illness in connection with the decentralization of the psychiatric treatment which has taken place in the Western world during the last 30-40 years (8).

Meta-analyses describe increased physical morbidity among patients with psychiatric diseases and increased mortality on account of somatic diseases (7). One of the reasons for the increased mortality could be the use of second generation antipsychotics that in some cases cause weight gain and metabolic syndrome which is associated with a two to threefold increase in cardiovascular mortality and a twofold increase in all-cause mortality (3;9). These effects would be expected to contribute to even higher mortality in the following years (10).

The use of more than one antipsychotic drug, polypharmacy, might also play a role (11;12). Psychiatric societies, national and international health authorities advise against the use of polypharmacy (13).

The quality of the general health care in patients with severe mental illness and the consensus about the prevention of somatic illness in this group of vulnerable patients need to be improved and there is evidence signifying the importance of the situation (14;15).

We need more knowledge about how to integrate the prevention and care of somatic illness to this group of patients with severe psychiatric illness.

This study investigates ways to improve the physical health of people with a psychiatric diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Living in one of the 6 institutions in Region Nordjylland

Exclusion Criteria:

* Not capable of speaking Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
waist circumferences | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mr Hjorth, MPH, Principal Investigator — Unit for Psychiatric research North Jutland; Povl Mr Munk Joergensen, Professor, Study Director — Unit for psychiatric research North Jutland
Locations (1):
- Enheden for psykiatrisk forskning, Aalborg, Denmark